CLINICAL TRIAL: NCT03859596
Title: Revisional Surgery After 925 OAGB Operations Retrospective Cohort Study of the United Kingdom MGB[Mini Gastric Bypass]/OAGB Collaborative Group.
Brief Title: Revisional Surgery After 925 OAGB[One Anastomosis Gastric Bypass] Operations Retrospective Cohort Study of the UK MGB/OAGB Collaborative Group.
Status: Completed | Type: Observational
Sponsor: ABDULZAHRA HUSSAIN (Other)
Collaborators: Phoenix Healthcare Group (Industry); Heart of England NHS Trust (Other); The Whittington Hospital NHS Trust (Other Government); Doncaster And Bassetlaw Hospitals NHS Foundation Trust (Other); Spire, Inc. (Industry); King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor-Investigator, ABDULZAHRA HUSSAIN, Consultant Surgeon, ParkHill Hospital
Organization: ParkHill Hospital (Other)
Other Study IDs: 0000
Record Dates: First submitted 2019-02-26; First posted 2019-03-01 (Actual); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: Revisions After MGB/OAGB; Morbidities; Morality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MGB/OAGB: Consequent group of patients who underwent MGB/OAGB
  Interventions: Procedure: MGB/OAGB

INTERVENTIONS:
Procedure: MGB/OAGB — BARIATRIC PROCEDURE INVOLVED CREATION OF SLENDER GASTRIC POUCH OF 12-15CM IN LENGTH AND BILIO-PANCREATIC LIMB OF 150-200 CM

SUMMARY:
Background: One anastomosis Gastric Bypass/Mini Gastric Bypass (OAGB/MGB) is a new operation that provides comparable outcomes to the common bariatric procedures. Revisional surgery is still needed after a number of OAGB/MGB procedures. The aim of this study is to report the causes and management of these revisions.

Methods: From 2010 -2018, 925 OAGB/MGB operations were performed at 7 bariatric units across the United Kingdom and included in this retrospective cohort study. The data was retrospectively collected and analysed. The primary end point was identification of the causes and management of revisions. Follow up ranged from 6 months to 3 years.

Results: Twenty-two patients (2.3%) required revisional surgery after OAGB/MGB. Five patients (0.5%) developed severe diarrhoea managed by shortening the bilio-pancreatic limb (BPL) to 150cm. Four patients (0.4%) developed afferent loop syndrome and bile reflux was reported in another 3 (0.3%) cases; all were managed by either conversion to Roux en Y Gastric Bypass (RYGB) or a Braun anastomosis. Postoperative bleeding was controlled laparoscopically in 3 patients (0.3%). Liver decompensation was reported in 2 patients (0.2%) was treated by shortening the BPL in one patient and a reversal to normal anatomy in another. The liver failure resolved in both patients. Other indications for revision included two gastro-jejunal stenosis (0.2%), one perforated ulcer (0.1%), one patient (0.1%) with excessive weight loss and one case (0.1%) of protein malnutrition. None of the 22 patients undergoing revisional surgery after OAGB/MBG died. Lost to follow up rate was 0.2%.

Conclusion: Complications requiring revisional surgery after OAGB/MGB are uncommon (2.3%) and the majority can be managed by bilio-pancreatic limb shortening, the addition of a Braun side-to-side anastomosis or conversion to RYGB. Bilio-pancreatic limb length of 200 cm or more resulted in serious complications of liver failure, protein malnutrition, excessive weight loss and diarrhoea.

DETAILED DESCRIPTION:
The UK OAGB/MGB collaborative group of 12 consultant bariatric surgeons was founded in 2017 and the data of 925 OAGB/MGB procedures were retrospectively collected and analysed in this cohort study. The treatment pathway is the SAME at each NHS centre. The indications for referral, consultations, and follow up after surgery are similar. This is agreed bariatric practice governed by British Obesity and Metabolic Surgery Society's [BOMSS] guidance.

The patients' age, BMI, presence of T2DM, comorbidities, Gastro-oesophageal reflux and hiatus hernia, Barrett's oesophagus, family history of upper gastro-intestinal cancer, and the patient choice were the main factors to influence the decision to the procedure type. Each centre is offering Roux en Y Gastric Bypass (RYGB), Laparoscopic Sleeve Gastrectomy (LSG), MGB/OAGB and Adjustable Gastric Band (AGB). The allocation of the procedure is finalised after mutual agreement between the patient and the surgeon taking in consideration the above factors and patient's choice. The data was retrospectively collected by the surgical team at each institution and sent to the lead of the collaborative group. The follow up is conducted by clinical visits, blood tests and radiology [ultrasound, computed tomography ] when needed.

The procedures were performed between September 2010 and May 2018. A long gastric pouch of average 15cm was constructed over a 34-36F bougie using laparoscopic staplers. The start point of stapling is at the crow's foot. The omentum was only divided in selected cases such as male patients with a very high Body Mass Index (BMI). After identifying the duodeno-jejunal junction, a BPL ranging from 150-300 cm was measured. The end-side /side-side gastro-jejunostomy was made using a combined hand-sewn /stapled technique. Use of drains and closure of Petersen's space varied between different surgeons. The patients were discharged after 2-3 nights. The follow up was ranged from 6 months to 3 years. In the UK the NHS and private practice are following National Institute of Clinical Excellence [NICE] guidelines in management and post operative follow up. Thus there is very strict follow up for two years after the operation. The patients are seen two weeks after the primary surgery at which clinical examination, dietary assessment and baseline post operative blood test is performed. Then the patients are seen one month after that, then 3 monthly period for the initial year, and 6 monthly for the last year. During all these visits, clinical, dietary and routine biochemical assessments were conducted. For patients who developed complications, a different and longer pathway of follow up is adopted until they recover and then, discharged to their general practitioners (GPs). The paper was written to comply with STROCSS guidelines (www.strocssguideline.com).

ELIGIBILITY:
Inclusion Criteria:

1. They have a BMI of 40 kg/m2 or more, or between 35 kg/m2 and 40 kg/m2 and other significant disease (for example, type 2 diabetes or high blood pressure) that could be improved if they lost weight.
2. All appropriate non-surgical measures have been tried but the person has not achieved or maintained adequate, clinically beneficial weight loss.
3. The person has been receiving or will receive intensive management in a tier 3 service.
4. The person is generally fit for anaesthesia and surgery.
5. The person commits to the need for long-term follow-up.
6. Age 18-71 years -

Exclusion Criteria:

1. Less than 18 or more than 71 years of age
2. Not fit for bariatric surgery
3. Psychiatric illness -

Ages: 18 Years to 71 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Consequent series of obese patients with BMI more than 35 for English patients and more than 30 for Asians with comorbidities
Sampling Method: Non-Probability Sample
Enrollment: 925 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Morbidities assessed by liver failure, protien malnutrition, diarrhea , bleeding, afferent loop syndrome,stomal ulcer,perforation, leak,infection | 3 years
  Liver failure, protien malnutrition, diarrhea , bleeding, afferent loop syndrome, stomal ulcer perforation,leak,infection.

SECONDARY OUTCOMES:
Mortality | 3 years
  Death after revision

IPD SHARING:
Plan to Share IPD: Undecided